CLINICAL TRIAL: NCT04922723
Title: A Study of Radiation/Temozolomide and Immunotherapy With Daratumumab to Improve Antitumor Efficacy in Glioblastoma (PRIDE).
Brief Title: Radiation/Temozolomide and Immunotherapy With Daratumumab to Improve Antitumor Efficacy in Glioblastoma
Acronym: PRIDE
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Sonikpreet Aulakh, Assistant Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2109412076; IND# Pending (Other: FDA)
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma
Keywords: Immunotherapy; Radiation/Temozolomide; Antitumor Efficacy
MeSH Terms: conditions — Glioblastoma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab (Experimental): Daratumumab, IV, 16 mg/KG -
  1 dose prior to surgery or biopsy; Weeks 1 - 8 = 1 dose weekly; Weeks 9 - 24 = 1 dose every other week; Weeks 25 onward (determined by disease progression) = 1 dose every 4 weeks
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered by IV infusion to subjects in combination with current therapeutic strategies of surgical resection followed by a course of Temozolomide and radiation therapy.
  Other Names: Darzalex

SUMMARY:
TMZ is a standard therapy for GBM. The study will demonstrate that Daratumumab can collaborate with TMZ to enhance the cytotoxicity against GBM cells. Collectively, the preclinical data along with existing in vivo studies by others provides the rationale for therapeutic targeting of CD38 in GBM and its microenvironment. Daratumumab is commercially available, is safe and well tolerated when combined with alkylating chemotherapy, radiation therapy and has attained therapeutic CSF levels. Thus, the addition of Daratumumab to the frontline treatment regimen of GBM can potentially have a significant clinical benefit. Approximately 16 subjects will be enrolled in this trial. Up to 6 will be enrolled in the phase I part and 10 to 13 in the phase II part to come up with a total of 16 patients with 2 phases combined.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is an aggressive brain cancer. Current therapeutic strategies include maximal safe surgical resection followed by course of Temozolomide (TMZ) and radiation therapy (RT). Despite trimodality treatment, recurrence remains inevitable. Our study will use Daratumumab, an anti-CD38 monoclonal antibody, in combination with TMZ and RT in newly diagnosed GBM patients. There is pre-clinical evidence suggesting Daratumumab is cytotoxic to GBM in a multimodal fashion, its safe when combined with chemotherapy & radiation therapy as well as has the potential to cross blood brain barrier.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have high radiological likelihood of GBM with plan for resection/biopsy for histologically confirmed GBM
* ECOG Performance status ≤ 2

  * Subjects must have normal organ and marrow function as defined below:
  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST (SGOT) ≤ 3 X institutional upper limit of normal
  * ALT (SGPT) ≤ 3 X institutional upper limit of normal
  * Serum Creatinine within normal institutional limits OR glomerular filtration rate (GFR) 60 mL/min/1.73 m2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m2
* The effects of Daratumumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Daratumumab and TMZ administration.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who received prior treatment for GBM.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Daratumumab and TMZ.
* BCG (Intravesical), Deferiprone, and Dipyrone are risk X category and should be avoided when Daratumumab is used. Chloramphenicol (Ophthalmic), promazine and Clozapine are in the risk category C and myelosuppression signs should be monitored when used in combination with Daratumumab.
* Avoid category Risk X drugs such as BCG (Intravesical), Deferiprone, Dipyrone, Natalizumab, Tacrolimus (Topical), Vaccines (Live) and Pimecrolimus concurrently with TMZ. Consider therapy modifications of category D drugs such as Baricitinib, Echinacea, Fingolimod, Leflunomide, Lenograstim, Lipegfilgrastim, Nivolumab, Palifermin, Roflumilast, Tofacitinib, Vaccines (Inactivated when used with TMZ. Monitor therapy for category risk C drugs such as Chloramphenicol (Ophthalmic), CloZAPine, Coccidioides immitis Skin Test, Denosumab, Ocrelizumab, Pidotimod, Promazine, Sipuleucel-T, Trastuzumab, and Valproate Products.
* Patients with uncontrolled intercurrent illness.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because there are no animal and human data to assess the risk of Daratumumab during pregnancy. On the other hand, TMZ is a category D drug where adverse events are observed in animal reproduction studies. May cause fetal harm when administered to pregnant females. Male and female patients should use effective contraception to avoid pregnancy while receiving temozolomide. May impair male fertility based on animal data).
* Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal.

  o Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is <50% of predicted normal.
* Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification.

  o Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.
* Clinically significant cardiac disease, including:

  * Myocardial infarction within 6 months before randomization, or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV).
  * Uncontrolled cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) rate of Daratumumab | Up to 6 weeks
  Rate of subjects that experience DLT. Subjects will be evaluated for DLTs after 6 doses of Daratumumab. If there is no DLT in the first 3 patients, the investigators will move forward to conduct the phase II clinical trial. If there is a DLT, another three patients will be enrolled. The study may be suspended with additional discussions in the data monitoring committee if there are ≥2 identified DLTs in the first 3 patients or ≥2 DLTs in the first 6 patients. The sample size justification is based on the standard 3+3 design.
Phase II - Median overall survival of newly diagnosed GBM patients | Up to 12 months
  Evaluate the median overall survival of newly diagnosed GBM patients. All patients in phase I part will be included in the efficacy analysis on overall survival (OS) in phase II part. If the 1-year survival rate of the study subjects is above 50% (median survival rate), it will be considered that the new intervention is promising.

SECONDARY OUTCOMES:
Phase I - Median overall survival of newly diagnosed GBM patients | Up to 6 weeks
  Evaluate the median overall survival of newly diagnosed GBM patients. All patients in phase I part will be included in the efficacy analysis on overall survival (OS) in phase II part. If the 1-year survival rate of the study subjects is above 50% (median survival rate), it will be considered that the new intervention is promising.
Phase I - Evaluate the Progression-Free Survival (PFS) | Up to 6 weeks
  Duration of time from start of Daratumumab treatment to time of progression or death, whichever occurs first.
Phase I - Assess the treatment-emergent adverse events | Up to 6 weeks
  Treatment-emergent Adverse Events are events not present prior to the initiation of treatment or any event already present that worsens in either intensity or frequency following the treatment.
Phase I - Estimate the tumor response rate | Up to 6 weeks
  To estimate tumor response rates after treatment with Daratumumab.
Phase II - Evaluate the Progression-Free Survival (PFS) | Up to 12 months
  Duration of time from start of Daratumumab treatment to time of progression or death, whichever occurs first.
Phase II - Assess the treatment-emergent adverse events | Up to 12 months
  Treatment-emergent Adverse Events are events not present prior to the initiation of treatment or any event already present that worsens in either intensity or frequency following the treatment.
Phase II - Estimate the tumor response rate | Up to 12 months
  To estimate tumor response rates after treatment with Daratumumab.

CONTACTS AND LOCATIONS:
Overall Officials: Sonikpreet Aulakh, MD, Principal Investigator — WVU Cancer Institute
Locations (1):
- West Virginia University Cancer Institute Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No